CLINICAL TRIAL: NCT02083991
Title: A Controlled Randomized, Open-label, Multi-centre Study Evaluating if a Steroid-free Immunosuppressive Protocol, Based ATG-induction, Low Tacrolimus-dose and Therapeutic Drug Monitoring of Mycophenolate Mofetil, Reduces the Incidence of New Onset Diabetes After Transplantations, in Comparison With Standard Steroid-based Protocol With Low-dose Tacrolimus.
Brief Title: Trial of Steroid Avoidance and Low-dose CNI by ATG-induction in Renal Transplantation
Acronym: SAILOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-000451-13
Record Dates: First submitted 2014-03-03; First posted 2014-03-11 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus
Keywords: NODAT; Renal transplantation; Corticosteroids avoidance; CNI minimization
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Steroid-free low TAC-arm (Experimental): Induction therapy: Thymoglobulin i.v. 2,5 mg/kg day 0 and 1, preceded by methylprednisolone i.v. 250 mg day 0 and 50 mg day 1.
  Maintenance therapy: Advagraf(TAC) 0,2 mg/kg p.o. started day1 (target concentration 5-10 ng/ml, after 3 months 4-7 ng/ml; MMF 1g x 2 p.o. (target Area Under Curve, AUC 40-60 mg.h/L); No steroids p.o.
  Interventions: Drug: Steroid-free low TAC-arm: Thymoglobulin Standard low-TAC arm: Simulect, prednisolon
- Standard low-TAC arm (Active Comparator): Induction therapy: Simulect i.v. 20 mg day 0 and 4; Steroids i.v. according to local practice.
  Maintenance therapy: Advagraf(TAC) p.o. 0,2 mg/(target concentration 5-10 ng/ml, after 3 months 4-7 ng/ml); MMF 1g x 2 p.o. (target AUC 40-60 mg.h/L); Steroids p.o. according to hospital practice (but not less than 5mg daily after 6 months).
  Interventions: Drug: Steroid-free low TAC-arm: Thymoglobulin Standard low-TAC arm: Simulect, prednisolon

INTERVENTIONS:
Drug: Steroid-free low TAC-arm: Thymoglobulin Standard low-TAC arm: Simulect, prednisolon

SUMMARY:
Balancing immunosuppressive treatment in organ transplantation in order to achieve effective prevention of rejection on one side and avoidance of negative side effects on the other side is a major challenge, leading to developing different immunosuppressive protocols. Cornerstones of immunosuppressive treatment such as Corticosteroids (CS) and Calcineurin Inhibitors (CNI) are known to cause an increased incidence of diabetes, cardiovascular morbidity, nephrotoxicity and malignancies.

The investigators believe that both avoidance of CS and minimization of CNI, while using Anti-ThymocyteGlobuline(ATG) induction (instead of interleucin-2 receptor blockers) and mycofenolate mofetil(MMF) therapeutic drug monitoring is going to reduce negative side effects, without increased rejection frequency in renal transplanted patients.

ELIGIBILITY:
Inclusion Criteria:

* First or second single kidney (cadaveric or living donors) transplant recipients.
* Considered for a standard immunosuppressive protocol.
* Must be capable of giving written informed connect for participation in the study for 24 months.

Exclusion Criteria:

* Diabetes mellitus or plasma glucose >11,1 at admission.
* Receiving steroids at the time of transplantation or likely to need steroids after transplantation.
* Multiorgan transplants and/or previously transplanted with any other organ than kidney.
* Panel reacting antibodies(PRA) >25% in most recent test or considered to be of high risk for rejection which requires an enhanced immunosuppression.
* Renal transplants from HLA-identical sibling.
* Hypersensitivity to, or disability to take immunosuppressive drugs.
* Blood group(ABO)-incompatible transplants.
* Unlikely to comply with the study requirements.
* Transplant from donor positive for HIV, HBsAg, Hepatitis C.
* Female of childbearing potential planing/being pregnant or unwilling to use contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of New Onset of Diabetes After Transplantation(NODAT) | 12 month after transplantation

SECONDARY OUTCOMES:
Cumulative incidence of NODAT | 3, 6, 24 month after transplantation
Composite measure | 12, 24 months
  Freedom from acute rejection, graft and patient survival
Renal function | 12, 24 months
  Evaluated by measured glomerular filtration rate (mGFR)
Incidence of acute rejection and chronic changes | 12 months
  Analysed by protocol biopsies, evaluated by the Banff system.
Incidence of hypertension | 3, 12, 24 months
  Standardized measurement.
Antihypertensive treatment | 3, 12, 24 months
  Number and type of antihypertensive drugs.
Lipid lowering drugs | 12, 24 months
  Number and type of lipid lowering drugs.
Incidence of antibody-mediated rejection | 12, 24 months
  Analysed by biopsies, evaluated by the Banff system, and by donor-specific HLA antibodies
Cumulative frequency of cardiovascular complications and events. | 10 days, 3, 12, 24 months
  Collecting Adverse Events (AE) reports
Cumulative frequency of malignancy. | 6, 12, 24 months
  Collecting AE reports
Cumulative frequency of infections | 10 days, 3, 6, 12, 24 months
  Collecting AE reports

CONTACTS AND LOCATIONS:
Overall Officials: Per Lindnér, MD, Principal Investigator — Transplant Center, Sahlgrenska University Hospital, Gothenburg, Sweden
Locations (1):
- Transplant Institute, Sahlgrenska University Hospital, Gothenburg, Sweden